CLINICAL TRIAL: NCT05448053
Title: Clinical and Radiographic Evaluation of Illizarov Fixation in Open Type III (A&B) Pediatric and Adolescent Tibial Shaft Fractures
Brief Title: Illizarov Fixation in Open Type III (A&B) Pediatric and Adolescent Tibial Shaft Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, khaled Gamal Amir, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Khaled381991
Record Dates: First submitted 2022-02-09; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-02

CONDITIONS: Open Type III (A&B)Pediatric and Adolescent Tibial Shaft Fractures; Ilizarov Fixation
MeSH Terms: interventions — Ilizarov Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ilizarov device (Experimental): Ilizarov fixation in open type III pediatric tibial shaft fractures
  Interventions: Procedure: Ilizarov

INTERVENTIONS:
Procedure: Ilizarov — Ilizarov fixation in open type III pediatric and adolescent tibial shaft fractures
  Other Names: ORIF with broad DCP

SUMMARY:
The Ilizarov method is our usual treatment of choice for open, complex, physeal or unstable fractures and for patients in whom non-operative or other treatments have failed .

DETAILED DESCRIPTION:
Tibial fractures are the third most common injury involving a long bone in children. Most occur in the distal third, and approximately 10% are open.High-energy injuries with soft tissue compromise or segmental bone loss, present specific challenges. There is a significant risk of nonunion (7.5%),malunion (17%),infection (10%),and loss of reduction (32%).Many forms of treatment are available including a cast, elastic nailing, and external fixation using either a monolateral fixator, or a circular frame . In complex adult tibial fractures, evidence for the effectiveness of definitive external fixation using a circular frame continues to emerge.Fixators may be used for the correction of tibial deformities in children.Currently, only relatively small case series have been published describing their use for trauma in children and adolescents, albeit with good results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 8-16 years old.
* Diagnosed to have open grade IIIA and IIIB tibial fracture according to Gustilo-Anderson fracture classification system.
* Fractures of the shaft of the tibia or distal tibial fractures involving the ankle joint and were complicated by bone and/or soft-tissue loss of more than 3 cm.
* An external fixator could be placed in the proximal lower extremity, distal lower extremity, or foot, and normal bone segments available for osteotomy.
* Admitted in the duration between 1st of January 2022 until end of December 2023.

Exclusion Criteria:

* Patients requiring free flap or local flap transfer to close the wound.
* Open grade IIIC tibial fractures (with vascular injury).
* Loss to follow-up.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Union of tibial fracture | 1 year
  Assess Union of the fracture using radiographic union scale in tibial fracture(RUST)

SECONDARY OUTCOMES:
Determine alignment | 1 year
  Determine alignment using slit scanogram for both Lower limbs
Patient reported outcome measures | 1 year
  Patient reported outcome measures using Stanmore limb reconstruction score (SLRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt